CLINICAL TRIAL: NCT05195502
Title: Cellular Composition of the Human Colon Using Single-cell RNA and Single-cell ATAC-sequencing.
Brief Title: Mapping the Human Colon Using Single Cell Sequencing
Acronym: COLATA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Bispebjerg Hospital (Other)
Collaborators: The Novo Nordisk Foundation Center for Basic Metabolic Research (Other)
Responsible Party: Principal Investigator, Jacob Antonsen, Senior Registrar, Bispebjerg Hospital
Other Study IDs: COLKEND01
Record Dates: First submitted 2022-01-07; First posted 2022-01-19 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2022-08

CONDITIONS: Diabetes; Large Bowel Cancer; Inflammatory Bowel Diseases
MeSH Terms: conditions — Diabetes Mellitus; Colonic Neoplasms; Inflammatory Bowel Diseases | interventions — Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1. Bloodsamples, including full blood, serum and plasma
  2. Endoscopic mucosal biopsies from the large bowel
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Screening colonoscopy patients: Patients referred for out-patient colonoscopy in the Danish Colorectal Screening program
  Interventions: Diagnostic Test: Biopsy

INTERVENTIONS:
Diagnostic Test: Biopsy — Participants included in the study, will have additional biopsies performed during their colonoscopy

SUMMARY:
The overall purpose of this study is to describe the cellular composition of the human colon and its gene expression using scRNAseq and scATACseq methods. This will potentially provide is with a detailed map of the colon aiding our understanding of how diseases of the colon develop as well as the colons influence on systemic diseases such as type II diabetes.

DETAILED DESCRIPTION:
The human colon is composed of four distinct histological layers: Serosa, muscularis externa, submucosa, and mucosa. The inner mucosal surface is composed of columnar epithelium and glandular tissue containing crypts of Lieberkühn and secretory goblet cells, lamina propria and muscularis mucosa. Several distinct cell types have been discovered in varying degree in the colon for example enteroendocrine cells and M-cells.

The cellular composition, patterns of gene expression and upstream regulatory pathways of the human colon varies across different anatomical location. This is evident in the anatomical bias in benign and malignant colorectal diseases. For example, the distal colon has a higher incidens of ulcerative colitis, diverticulitis, and chromosomal instability cancer whereas in the proximal colon ischemic colitis, collagenous colitis and microsatellite instability-induced cancer are predominant.

Currently there are no studies describing baseline data for genome-wide coding, methylation or gene expression related to specific anatomic locations in the human colon.

By using scRNAseq and scATACseq (Single-cell Assay of Transposase Accessible Chromatin sequencing) we will be able to map open regions in the cell's DNA and RNA, thus providing us with a unique "map" of the cells in the colon as well is their gene expression. ScATACseq visualizes open regions in the chromatin, generating "peaks" which can then be used to map DNA motifs, such as transcription factor binding sites. With the emergence of scATACseq, chromatin accessibility is in combination with gene expression data an extremely useful resource to study cell type specific regulatory DNA interactions. To further study the immunological aspects of the colon, we will extract immune cells from the colon. Lastly, full blood will be extracted to better analyze metabolic risk factors in relation to the colon's metabolic cellular regulation.

The overall purpose of this study is to describe the cellular composition of the human colon and its gene expression using scRNAseq and scATACseq methods. This will potentially provide is with a detailed map of the colon aiding our understanding of how diseases of the colon develop as well as the colons influence on systemic diseases such as type II diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for out-patient colonoscopy as a result of positive hemoccult.
* Patients able to read and understand danish.
* Patients able to give informed consent.
* Patients of Scandinavian ethnicity.

Exclusion Criteria:

* Previous large bowel resections
* Suspicion pre or intraoperatively of benign or malignant disease of the colon
* Known inflammatory bowel disease.
* Immuno-modulation treatment
* Chemotherapy.
* Daily smoking
* > 21 weekly units of alcohol
* < 18 years of age

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Citizens aged 50 to 74 are invited to partake in screening for bowel cancer every second year. Patients who accept referral based on a positive fecal immunochemical test, will be invited to participate in this study
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Profiling of open chromatin regions | 2 years
  Mapping of cell types, including rare cell types, using profiling of open chromatin regions. (ATAC-seq) in mucosal biopsies from the large bowel
Evaluation of metabolic profile | 2 years
  Using bioimpedance, insulin and glucose measurements and CHiP-seq we will determine patient phenotype and epigenetics to evaluate their metabolic risk-profile and correlate this to cell types in the large bowel

SECONDARY OUTCOMES:
Colonic biofilm | 2 years
  By sequencing bacterial DNA in our samples, we will evaluate the mucosa-associated microbiome of the large bowel. This will be correlated to the two primary outcome measures

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Antonsen, MD, Principal Investigator — Bispebjerg Hospital
Locations (1):
- Bispebjerg University Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
Data in this study is based on biological samples and data from patient registry. These data are protected by the Danish Act on Processing of Personal Data and can be accessed through application to and approval from the Danish Data Protection Agency and the Danish Health Data Authority [https://sundhedsda tastyrelsen.dk/da/forskerservice/ansog-om-data] where the purpose and the feasibility of the intended analysis should be accounted for.

REFERENCES:
- [Background] Kaz AM, Wong CJ, Dzieciatkowski S, Luo Y, Schoen RE, Grady WM. Patterns of DNA methylation in the normal colon vary by anatomical location, gender, and age. Epigenetics. 2014 Apr;9(4):492-502. doi: 10.4161/epi.27650. Epub 2014 Jan 10. PMID 24413027
- [Background] Knight JM, Kim E, Ivanov I, Davidson LA, Goldsby JS, Hullar MA, Randolph TW, Kaz AM, Levy L, Lampe JW, Chapkin RS. Comprehensive site-specific whole genome profiling of stromal and epithelial colonic gene signatures in human sigmoid colon and rectal tissue. Physiol Genomics. 2016 Sep 1;48(9):651-9. doi: 10.1152/physiolgenomics.00023.2016. Epub 2016 Jul 8. PMID 27401218
- [Background] Forgue-Lafitte ME, Fabiani B, Levy PP, Maurin N, Flejou JF, Bara J. Abnormal expression of M1/MUC5AC mucin in distal colon of patients with diverticulitis, ulcerative colitis and cancer. Int J Cancer. 2007 Oct 1;121(7):1543-9. doi: 10.1002/ijc.22865. PMID 17565737
- [Background] Costales-Carrera A, Fernandez-Barral A, Bustamante-Madrid P, Dominguez O, Guerra-Pastrian L, Cantero R, Del Peso L, Burgos A, Barbachano A, Munoz A. Comparative Study of Organoids from Patient-Derived Normal and Tumor Colon and Rectal Tissue. Cancers (Basel). 2020 Aug 15;12(8):2302. doi: 10.3390/cancers12082302. PMID 32824266
- [Background] Buenrostro JD, Wu B, Chang HY, Greenleaf WJ. ATAC-seq: A Method for Assaying Chromatin Accessibility Genome-Wide. Curr Protoc Mol Biol. 2015 Jan 5;109:21.29.1-21.29.9. doi: 10.1002/0471142727.mb2129s109. PMID 25559105